CLINICAL TRIAL: NCT01245140
Title: Efficacy of Oral Alitretinoin Treatment in Patients With Palmo-plantar Pustulosis (PPP) Inadequately Responding to Standard Topical Treatment
Brief Title: Efficacy of Alitretinoin Treatment in Patients With Pustular Form of Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 117221; 2010-022843-39 (EudraCT Number); BAP02028 (Other: Basilea Pharmecutica)
Record Dates: First submitted 2010-11-16; First posted 2010-11-22 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-12-21 (Actual); Status verified 2017-11

CONDITIONS: Psoriasis
Keywords: Palmo-Plantar Pustolosis
MeSH Terms: conditions — Psoriasis | interventions — Alitretinoin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Active Comparator): to receive study drug (alitretinoin, 20 patients)
  Interventions: Drug: alitretinoin
- Placebo (Placebo Comparator): to receive placebo (dummy drug, 10 patients)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: alitretinoin — to receive verum (20 patients)
  Other Names: Toctino
  Arms: Active
Drug: Placebo — to receive placebo (10 patients)
  Arms: Placebo

SUMMARY:
The main purpose of this study is to demonstrate the improvement in the skin condition rate of patients receiving alitretinoin compared to patients receiving placebo.

DETAILED DESCRIPTION:
Palmo-plantar pustulosis (PPP) is an inflammatory skin disease affecting palms and soles. The disease is considered as a sub-form of psoriasis and presents with sterile pustules of the palms and the soles. This study investigates the efficacy of alitretinoin in patients who have not responded to topical drugs (e.g., steroid creams), who are suffering for at least 6 month from the condition and whose disease severity is confirmed by a score.

ELIGIBILITY:
Inclusion Criteria:

1. A female subject is eligible to participate if she is of:

   * Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea and a follicle stimulating hormone concentration of ≥40 international units (IU)/L.
   * Child-bearing potential with negative pregnancy test as determined by human chorionic gonadotropin (hCG) test at screening or prior to dosing and either 1) agrees to use a medically acceptable contraception method for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point and continue contraception until the end of the study, or 2) has only same-sex partners, when this is her preferred and usual lifestyle.
2. Capable of understanding and willing to provide signed and dated written voluntary informed consent (and any local or national authorization requirements) before any protocol specific procedures are performed.
3. Male or female aged at least 18 years at time of consent and at time of first dose.
4. Have PPP for at least 6 months, with or without psoriasis lesions on other areas of the skin
5. A PPPASI score of at least 8 with involvement of at least 10% of the palms and/or the soles
6. Refractory to standard topical corticosteroid therapy

Exclusion Criteria:

1. Unable to comply with the requirement of the study
2. Female subjects who are pregnant or who plan to become pregnant or who are breast feeding
3. Subjects whose disease is adequately controlled by standard non-medicated therapy (skin moisturizing and protection)
4. Known hypersensitivity to other retinoids or vitamin A derivatives, or to any study medication component, especially soybean oil and partly hydrogenated soybean oil
5. Treated with any of the following treatments 4 weeks before the start of study treatment:

   * systemic drugs: corticosteroids, immunosuppressants, methotrexate
   * phototherapy: ultraviolet B light therapy [UVB], psoralen with ultraviolet A combination therapy [PUVA], Grenz rays, X-rays
6. Treated with biologic treatments within 6 weeks prior to start of study treatment.
7. Abnormal hematology
8. Treated with any systemic or topical retinoids within 3 months or 1 month, respectively, before start of study treatment
9. Treated with high-potency topical corticosteroids within 2 weeks before the start of study treatment
10. Severe generalized pustular psoriasis
11. A skin condition of palms and/or soles that interferes with the diagnosis of PPP by the investigator
12. Any condition that, in the judgment of the investigator, would put the subject at unacceptable risk for participation in the study.
13. Hepatic insufficiency, severe renal failure, uncontrolled hypercholesterolemia as characterized by:

    * AST/ ALT >2.5 x upper limit of normal (ULN)
    * Creatinine clearance <60 mL/min (calculated, Cockcroft-Gault)
    * Fasting triglyceridemia >1.5 x upper limit of normal (ULN)
    * Fasting cholesterol >1.5 x ULN
    * Fasting low-density lipoprotein (LDL) cholesterol >1.5x ULN
14. Subjects with hypothyroidism as indicated by thyroid stimulating hormone (TSH) above ULN and thyroxine (T4) test below LLN or hypervitaminosis A
15. Subjects with unstable cardiac disease or poorly controlled cardiovascular risk factors, for example:

    * Acute coronary syndrome or coronary revascularization (percutaneous coronary intervention [PCI], coronary artery bypass graft [CABG]) within 3 months before start of study treatment
    * Poorly controlled diabetes mellitus (HbA1c >8.5%)
16. Systolic blood pressure ≥160 mm Hg and/or diastolic blood pressure ≥100 mm Hg at the screening examination
17. Subjects receiving drugs with a potential for drug-drug interaction, such as systemic tetracyclines, ketoconazole, or St. John's Wort within 1 week, or receiving systemic itraconazole within 2 weeks, before start of study treatment
18. Subjects included in the study of an investigational drug within 2 months before start of study treatment (3 months for biologics)
19. Subjects with a score of 20 or more on the Center for Epidemiologic Studies Depression scale (CES-D), or with active major psychiatric disorder (eg, Major Depressive Disorder, Generalized Anxiety Disorder, Bipolar Disorder [I or II], or schizophrenia)
20. Subjects who score a 4 or 5 for the previous 30 days on the Columbia Suicide Severity Rating Scale (CSSRS) at Screening or Baseline
21. Subjects who have made a suicide attempt within the 6 months preceding the Screening or Baseline visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-04-26 (Actual); Primary Completion 2014-03-12 (Actual); Study Completion 2014-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- GSK Investigational Site, Paris, France
- Germany (4):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Witten, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- GSK Investigational Site, Nijmegen, Netherlands
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 117221 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 117221 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 117221 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 117221 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 117221 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 117221 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 117221 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 7 centers from 26 April 2011 to 16 April 2014, in male and female participants of Palmo-plantar pustulosis (PPP), aged >= 18 years.
Pre-assignment Details: The total study duration was 33 weeks, with a Screening Period of up to 4 weeks, followed by 24 weeks of treatment and a 5-week safety Follow-up Period. Participants who met eligibility criteria were randomized (2:1) to receive 30 milligrams (mg) alitretinoin or matching placebo, given orally as gelatin capsules, once daily (QD) for up to 24 weeks.
Groups:
- Matching Placebo: Participants received matching placebo orally once daily (QD) for up to 24 weeks.
- Alitretinoin 30 mg: Participants received an alitretinoin 30 milligram (mg) capsule orally QD for up to 24 weeks.
Period: Overall Study
Arm/Group | Matching Placebo | Alitretinoin 30 mg
Started | 9 | 24
Completed | 6 | 14
Not Completed | 3 | 10
Not completed — Adverse Event | 1 | 3
Not completed — Lack of Efficacy | 2 | 4
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Refused Treatment/Did Not Coopera | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Matching Placebo: Participants received matching placebo orally QD for up to 24 weeks.
- Alitretinoin 30 mg: Participants received an alitretinoin 30 mg capsule orally QD for up to 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Matching Placebo | Alitretinoin 30 mg | Total
Number analyzed (Participants) | 9 | 24 | 33
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.00 (16.32) | 48.83 (14.94) | 48.88 (15.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 14 | 19
  Male | 4 | 10 | 14
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian/White | 8 | 22 | 30
  Oriental | 1 | 0 | 1
  Black | 0 | 1 | 1
  North African | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Palmo-plantar Pustulosis Psoriasis Area and Severity Index (PPPASI) Score at the End of Treatment (EOT) (Week 24) or at the Last Assessment
Description: The investigator evaluated the PPPASI score on a 5-point scale. The parameters of erythema, total number of pustules, and desquamation were scored for the right/left palm and the right/left sole. After correcting the scores for area (based on a 7-point scale) and the site involved (palm or sole), the PPPASI score per palm/sole was produced. The final PPPASI score was calculated as the sum of the PPPASI score for the right sole + the PPPASI score for the left sole + the PPPASI score for the right palm + the PPPASI score for the left palm and ranges from 0 (no palmo-plantar pustulosis psoriasis [PPP]) to 72 (most severe PPP). Change from Baseline is defined as value at the EOT minus the Baseline value.
Time Frame: Baseline and EOT (Week 24) or the last assessment
Population: Full Analysis Set : treated participants with >=1 efficacy result after receiving study medication.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Matching Placebo | Alitretinoin 30 mg
Number analyzed (Participants) | 9 | 22
Scores on a scale | -44.6 (45.9) | -45.2 (32.8)
Statistical Analysis 1: Comparison: Matching Placebo vs Alitretinoin 30 mg; Test type: Superiority or Other; p = 0.9705, ANCOVA; Mean Difference (Net) = 0.5731, 95% CI 2-sided [-30.9738 to 32.1200]

2. Primary Outcome: Number of Participants With PPPASI 50 Response and PPPASI 75 Response
Description: The investigator evaluated the PPPASI score on a 5-point scale. The parameters of erythema, total number of pustules, and desquamation were scored for the right/left palm and the right/left sole. After correcting the scores for area (based on a 7-point scale) and the site involved (palm or sole), the PPPASI score per palm/sole was produced. The final PPPASI score was calculated as the sum of the PPPASI score for the right sole + the PPPASI score for the left sole + the PPPASI score for the right palm + the PPPASI score for the left palm and ranges from 0 (no palmo-plantar pustulosis psoriasis [PPP]) to 72 (most severe PPP). Change from Baseline is defined as value at the EOT minus the Baseline value. PPPASI 50 response and PPPASI 75 response are defined as a 50% and 75% decrease, respectively, in the PPPASI score from Baseline.
Time Frame: From Baseline until EOT (Week 24) or the last assessment
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Matching Placebo | Alitretinoin 30 mg
Number analyzed (Participants) | 9 | 22
Participants
  PPPASI 50 response | 6 | 11
  PPPASI 75 response | 3 | 5
Statistical Analysis 1: Comparison: Matching Placebo vs Alitretinoin 30 mg; Test type: Superiority or Other; p = 0.4564, Fisher Exact — PPPASI 50 response
Statistical Analysis 2: Comparison: Matching Placebo vs Alitretinoin 30 mg; Test type: Superiority or Other; p = 0.6595, Fisher Exact — PPPASI 75 response

3. Secondary Outcome: Total Pustule Count at Baseline; Weeks 4, 8, 12, 16, and 20; and at EOT (Week 24)
Description: The overall number of fresh and older pustules on the left and right palms and soles was assessed at Baseline, at each visit during the treatment period (Weeks 4, 8, 12, 16, and 20), and at the EOT visit. The total pustule count was calculated as the sum of the pustule count for the left/right palm and left/right sole.
Time Frame: Baseline; Weeks 4, 8, 12, 16, and 20; and EOT (Week 24)
Population: Full Analysis Set. Only participants available at the specified time points were analyzed (n=X, X).
Measure: Mean (Standard Deviation); unit: Pustule count
Arm/Group | Matching Placebo | Alitretinoin 30 mg
Number analyzed (Participants) | 9 | 22
Pustule count
  Baseline, n=9, 22 | 82.7 (59.1) | 106.0 (128.2)
  Week 4, n=9, 20 | 71.6 (66.5) | 31.0 (43.5)
  Week 8, n=7, 20 | 69.7 (30.8) | 30.4 (38.6)
  Week 12, n=7, 17 | 70.4 (63.2) | 21.5 (37.8)
  Week 16, n=6, 16 | 26.8 (25.5) | 26.0 (42.0)
  Week 20, n=6, 14 | 35.8 (37.7) | 30.5 (51.2)
  End of Treatment, n=8, 20 | 55.4 (104.5) | 33.6 (49.6)

4. Secondary Outcome: Absolute Change From Baseline (BL) in Total Pustule Count at Weeks 4, 8, 12, 16, and 20 and at EOT (Week 24)
Description: The overall number of fresh and older pustules on the left and right palms and soles was assessed at Baseline, at each visit during the treatment period (Weeks 4, 8, 12, 16, and 20), and at the End of Treatment visit. The total pustule count was calculated as the sum of the pustule count for the left/right palm and left/right sole. Change from Baseline is defined as the value at the post-Baseline visit minus the Baseline value.
Time Frame: Baseline; Weeks 4, 8, 12, 16, and 20; and EOT (Week 24)
Population: Full Analysis Set. Only participants available at the specified time points were analyzed (n=X, X).
Measure: Mean (Standard Deviation); unit: Pustule count
Arm/Group | Matching Placebo | Alitretinoin 30 mg
Number analyzed (Participants) | 9 | 22
Pustule count
  Week 4, n=9, 20 | -11.1 (58.4) | -75.3 (113.2)
  Week 8, n=7, 20 | -7.9 (51.5) | -75.9 (124.4)
  Week 12, n=7, 17 | -7.1 (75.5) | -74.2 (111.7)
  Week 16, n=6, 16 | -55.2 (56.5) | -75.6 (113.0)
  Week 20, n=6, 14 | -46.2 (37.8) | -65.1 (106.4)
  End of Treatment, n=8, 20 | -31.3 (79.4) | -82.1 (121.3)
Statistical Analysis 1: Comparison: Matching Placebo vs Alitretinoin 30 mg; Test type: Superiority or Other; p = 0.51, Wilcoxon test: Exact Test — Change in Total Pustule Count: BL to Last Visit

5. Secondary Outcome: Mean Modified Psoriasis Area Severity Index (mPASI) Score at Baseline; Weeks 4, 8, 12, 16, and 20; and EOT (Week 24)
Description: Psoriatic plaques were graded based on three criteria: redness (R), thickness (T), and scaliness (S). Severity was rated for each criterion on a 5-point scale (0=no involvement, up to 4=severe involvement). Fraction of the total surface area affected on the head, upper extremities, trunk, and lower extremities was graded on a 7-point scale (0=no involvement, up to 6=greater than 90% involvement). The four body regions were weighted to reflect their respective proportion of body surface area, and the composite mPASI score for all body regions was calculated based on the redness, thickness, and scaliness scores of plaques (0-4 each) for the head, upper extremities, trunk, and lower extremities and the area of psoriatic involvement score (0-6). The lowest possible mPASI score was zero and highest up to 72; Higher score values represents greater severity of psoriasis. mPASI scores were continuous, with 0.1 increments within these values.
Time Frame: Baseline; Weeks 4, 8, 12, 16, and 20; and EOT (Week 24)
Population: Full Analysis Set. Only participants available at the specified time points were analyzed (n=X, X).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Matching Placebo | Alitretinoin 30 mg
Number analyzed (Participants) | 9 | 22
Scores on a scale
  Baseline, n=9, 21 | 0.2 (0.4) | 0.5 (0.9)
  Week 4, n=9, 20 | 0.3 (0.6) | 0.4 (0.9)
  Week 8, n=7, 20 | 0.0 (0.1) | 0.4 (0.9)
  Week 12, n=7, 17 | 0.0 (0.1) | 0.4 (0.9)
  Week 16, n=6, 16 | 0.0 (0.0) | 0.2 (0.5)
  Week 20, n=6, 14 | 0.0 (0.1) | 0.1 (0.3)
  End of Treatment, n=8, 20 | 0.7 (1.9) | 0.3 (0.7)
Statistical Analysis 1: Comparison: Matching Placebo vs Alitretinoin 30 mg; Test type: Superiority or Other; p = 0.12, Wilcoxon test: Exact Test — Relative change in mPASI score: BL to Last Visit

6. Secondary Outcome: Change From Baseline in the mPASI Score at EOT (Week 24) or at the Last Assessment
Description: Psoriatic plaques were graded based on three criteria: redness (R), thickness (T), and scaliness (S). Severity was rated for each criterion on a 5-point scale (0=no involvement, up to 4=severe involvement). Fraction of the total surface area affected on the head, upper extremities, trunk, and lower extremities was graded on a 7-point scale (0=no involvement, up to 6=greater than 90% involvement). The four body regions were weighted to reflect their respective proportion of body surface area, and the composite mPASI score for all body regions was calculated based on redness, thickness, and scaliness scores of plaques (0-4 each) for head, upper extremities, trunk, lower extremities and area of psoriatic involvement score (0-6). Lowest possible mPASI score was 0 and highest up to 72; Higher score values represents greater severity of psoriasis. mPASI scores were continuous, with 0.1 increments within these values. Change from Baseline is defined as the value at EOT minus baseline value.
Time Frame: Baseline and EOT (Week 24) or the last assessment
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Matching Placebo | Alitretinoin 30 mg
Number analyzed (Participants) | 9 | 22
Scores on a scale | -95.8 (7.2) | -51.0 (38.3)
Statistical Analysis 1: Comparison: Matching Placebo vs Alitretinoin 30 mg; Test type: Superiority or Other; p = 0.2358, ANCOVA; Least squared estimation = 49.4927, 95% CI 2-sided [-49.0830 to 148.07]

7. Secondary Outcome: Number of Participants With mPASI 50 Response and mPASI 75 Response
Description: Psoriatic plaques were graded based on three criteria: redness (R), thickness (T), and scaliness (S). Severity was rated for each criterion on a 5-point scale (0=no involvement, up to 4=severe involvement). The fraction of the total surface area affected on the head, upper extremities, trunk, and lower extremities was graded on a 7-point scale (0=no involvement, up to 6=greater than 90% involvement). The four body regions were weighted to reflect their respective proportion of body surface area, and the composite mPASI score for all body regions was calculated. mPASI 50 response and mPASI 75 response is defined as a 50% and 75% decrease, respectively, in the mPASI score from Baseline.
Time Frame: From Baseline until EOT (Week 24)
Population: Full analysis set. Participants with lesions in areas of the body other than the hands and feet were assessed.
Measure: Number; unit: Participants
Arm/Group | Matching Placebo | Alitretinoin 30 mg
Number analyzed (Participants) | 3 | 6
Participants
  mPASI 50 response | 3 | 2
  mPASI 75 response | 3 | 2
Statistical Analysis 1: Comparison: Matching Placebo vs Alitretinoin 30 mg; Test type: Superiority or Other; p = 0.1667, Fisher Exact — mPASI 50 response
Statistical Analysis 2: Comparison: Matching Placebo vs Alitretinoin 30 mg; Test type: Superiority or Other; p = 0.1667, Fisher Exact — mPASI 75 response

8. Secondary Outcome: Mean Nail Psoriasis Severity Index (NAPSI) Score for Nail Bed Psoriasis and Nail Matrix Psoriasis at Baseline, Week 12, and EOT (Week 24)
Description: The severity of nail lesions was assessed for all participants with psoriatic nail involvement by obtaining the NAPSI score. Scores were taken for fingernails only. No scores were taken for participants with traumatic or fungal changes in nails. The nail was divided into four quadrants, each of which was rated with a 0 or 1, based on the absence (0) or presence (1) of pathological signs resulting from involvement of both the nail matrix and the nail bed. Each nail was given a score for nail bed psoriasis (0-4) and nail matrix psoriasis (0-4) depending on the presence of nail psoriasis in that quadrant. Possible scores for matrix and nail bed psoriasis: 0=none, 1=present in 1/4 nail, 2=present in 2/4 nail, 3=present in 3/4 nail, 4=present in 4/4 nail. NAPSI score for nail matrix (0-4) and nail bed (0-4) were reported at Baseline, Week 12, and at the EOT visit (Week 24).
Time Frame: Baseline, Week 12, and EOT (Week 24)
Population: Full Analysis Set. Only participants available at the specified time points were analyzed (n=X, X).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Matching Placebo | Alitretinoin 30 mg
Number analyzed (Participants) | 9 | 22
Scores on a scale
  NAPSI-bed, Baseline, n=9, 20 | 1.1 (2.3) | 1.2 (1.9)
  NAPSI-bed, Week 12, n=7, 17 | 0.4 (1.1) | 1.3 (3.3)
  NAPSI-bed, End of Treatment, n=8, 19 | 1.6 (2.8) | 0.9 (2.0)
  NAPSI-matrix, Baseline, n=9, 20 | 3.9 (6.2) | 3.6 (6.2)
  NAPSI-matrix, Week 12, n=7, 17 | 2.1 (3.7) | 2.6 (6.0)
  NAPSI-matrix, End of Treatment, n=8, 19 | 4.3 (6.0) | 2.6 (6.0)

9. Secondary Outcome: Absolute Change From Baseline in NAPSI Score for Nail Bed Psoriasis and Nail Matrix Psoriasis at Week 12, and EOT (Week 24)
Description: The severity of nail lesions was assessed for all participants with psoriatic nail involvement by obtaining the NAPSI score. Scores were taken for fingernails only. No scores were taken for participants with traumatic or fungal changes in nails. The nail was divided into four quadrants, each of which was rated with a 0 or 1, based on the absence (0) or presence (1) of pathological signs resulting from involvement of both the nail matrix and the nail bed. Each nail was given a score for nail bed psoriasis (0-4) and nail matrix psoriasis (0-4) depending on the presence of nail psoriasis in that quadrant. Possible scores for matrix and nail bed psoriasis: 0=none, 1=present in 1/4 nail, 2=present in 2/4 nail, 3=present in 3/4 nail, 4=present in 4/4 nail. NAPSI score for nail matrix (0-4) and nail bed (0-4) were reported at Baseline, Week 12, and at the EOT visit (Week 24). Change from Baseline is defined as the value at the post-Baseline visit minus the Baseline value.
Time Frame: Baseline, Week 12, and EOT (Week 24)
Population: Full Analysis Set. Only participants available at the specified time points were analyzed (n=X, X).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Matching Placebo | Alitretinoin 30 mg
Number analyzed (Participants) | 9 | 22
Scores on a scale
  NAPSI-bed, Week 12, n=7, 17 | -0.4 (1.1) | 0.3 (2.4)
  NAPSI-bed, End of Treatment, n=8, 18 | 0.4 (2.2) | -0.3 (1.6)
  NAPSI-matrix, Week 12, n=7, 17 | -1.4 (3.8) | -0.5 (2.0)
  NAPSI-matrix, End of Treatment, n=8, 18 | 0.8 (5.5) | -0.1 (5.0)

10. Secondary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE) and an AE/SAE Related to Study Treatment
Description: An AE was any adverse change from the participant's Baseline (pre-treatment) clinical condition, including intercurrent illness, which occurred during the course of a clinical study after written informed consent had been given, whether considered related to treatment or not. The relationship of AEs to the study treatment was assessed as unrelated, remotely related, possibly related, and probably related. For an AE to be considered serious, it fell into one or more of the following categories: results in death, is life threatening, results in persistent or significant disability/incapacity, results in or prolongs inpatient hospitalization, and is a congenital abnormality or birth defect.
Time Frame: From Baseline until safety follow up (Week 29)
Population: Safety Population: all randomized participants who received at least one dose of study medication
Measure: Number; unit: Participants
Arm/Group | Matching Placebo | Alitretinoin 30 mg
Number analyzed (Participants) | 9 | 24
Participants
  Any AE | 8 | 18
  Any AE remotely related to study medication | 6 | 15
  Any SAE | 0 | 1
  Any SAE remotely related to study medication | 0 | 1

11. Secondary Outcome: Absolute Change From Baseline in Fasted Lipid Laboratory Test Values at Weeks 4, 8, 12, 16, and 20; EOT (Week 24); and at Safety Follow-up (Week 29)
Description: Fasted lipid laboratory parameters included triglycerides, total cholesterol, high-density lipoprotein (HDL) cholesterol, and low-density lipoprotein (LDL) cholesterol. Change from Baseline is defined as the value at the post-Baseline visit minus the Baseline value.
Time Frame: Baseline; Weeks 4, 8, 12, 16, and 20; EOT (Week 24); and safety follow-up (Week 29)
Population: Safety Population. Only participants available at the specified time points were analyzed (n=X, X).
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Matching Placebo | Alitretinoin 30 mg
Number analyzed (Participants) | 9 | 24
Millimoles per liter (mmol/L)
  Triglycerides, Week 4, n=9, 19 | 0.6 (2.3) | 2.4 (3.7)
  Triglycerides, Week 8, n=7, 20 | 1.0 (1.9) | 3.8 (5.7)
  Triglycerides, Week 12, n=6, 17 | 2.5 (3.6) | 5.8 (8.7)
  Triglycerides, Week 16, n=5, 16 | 2.6 (1.7) | 4.2 (5.2)
  Triglycerides, Week 20, n=6, 14 | 2.6 (4.1) | 5.6 (6.2)
  Triglycerides, End of Treatment, n=7, 20 | -0.7 (2.5) | 3.3 (5.6)
  Triglycerides, safety follow-up, n=9, 21 | 1.2 (3.4) | 2.8 (5.8)
  Total cholesterol, Week 4, n=9, 19 | 0.0 (0.5) | 0.6 (0.6)
  Total cholesterol, Week 8, n=7, 20 | -0.2 (0.5) | 0.7 (0.8)
  Total cholesterol, Week 12, n=6, 17 | 0.1 (0.3) | 0.7 (0.9)
  Total cholesterol, Week 16, n=5, 16 | 0.1 (0.5) | 0.6 (0.8)
  Total cholesterol, Week 20, n=6, 14 | 0.1 (0.8) | 0.7 (1.1)
  Total cholesterol, End of Treatment, n=8, 20 | -0.1 (0.5) | 0.7 (0.7)
  Total cholesterol, safety follow-up, n=9, 22 | -0.0 (0.5) | 0.3 (0.8)
  HDL cholesterol, Week 4, n=8, 19 | -0.1 (0.2) | -0.1 (0.1)
  HDL cholesterol, Week 8, n=7, 20 | -0.1 (0.2) | -0.2 (0.2)
  HDL cholesterol, Week 12, n=6, 17 | -0.0 (0.2) | -0.2 (0.2)
  HDL cholesterol, Week 16, n=5, 16 | -0.1 (0.1) | -0.2 (0.2)
  HDL cholesterol, Week 20, n=6, 14 | -0.0 (0.2) | -0.2 (0.2)
  HDL cholesterol, End of Treatment, n=7, 20 | -0.1 (0.2) | -0.1 (0.2)
  HDL cholesterol, safety follow-up, n=9, 22 | -0.1 (0.2) | -0.0 (0.2)
  LDL cholesterol, Week 4, n=8, 19 | 0.2 (0.3) | 0.6 (0.5)
  LDL cholesterol, Week 8, n=7, 20 | 0.0 (0.5) | 0.5 (0.6)
  LDL cholesterol, Week 12, n=6, 17 | -0.1 (0.4) | 0.6 (0.6)
  LDL cholesterol, Week 16, n=5, 16 | 0.0 (0.5) | 0.4 (0.5)
  LDL cholesterol, Week 20, n=6, 14 | -0.0 (0.6) | 0.6 (0.9)
  LDL cholesterol, End of Treatment, n=7, 20 | 0.0 (0.4) | 0.4 (0.6)
  LDL cholesterol, safety follow-up, n=9, 22 | 0.0 (0.3) | 0.3 (0.5)

12. Secondary Outcome: Absolute Change From Baseline in Fasted LDL/HDL Ratio at Weeks 4, 8, 12, 16, and 20; EOT (Week 24); and at Safety Follow-up (Week 29)
Description: Change from Baseline is defined as the value at the safety follow up visit minus baseline value.
Time Frame: Baseline; Weeks 4, 8, 12, 16, and 20; EOT (Week 24) and safety follow-up (Week 29)
Population: Safety Population. Only participants available at the specified time points were analyzed (n=X, X).
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Matching Placebo | Alitretinoin 30 mg
Number analyzed (Participants) | 9 | 24
Ratio
  Baseline, n=7, 22 | 0.0 (0.0) | 0.0 (0.0)
  Week 4, n=6, 17 | 0.3 (0.2) | 0.7 (0.4)
  Week 8, n=6, 18 | 0.2 (0.6) | 0.9 (0.6)
  Week 12, n=5, 16 | 0.2 (0.4) | 0.9 (0.9)
  Week 16, n=5, 15 | 0.1 (0.5) | 0.9 (0.7)
  Week 20, n=6, 13 | 0.0 (0.5) | 0.7 (1.1)
  End of Treatment, n=7, 19 | 0.1 (0.4) | 0.5 (0.8)
  Safety follow-up, n=7, 20 | 0.1 (0.4) | 0.1 (0.6)

13. Secondary Outcome: Number of Participants With the Indicated Shift in the Indicated Laboratory Values From Baseline (BL) to EOT (Week 24)
Description: Laboratory parameters included triglycerides, total cholesterol, HDL cholesterol, LDL cholesterol, LDL/HDL ratio, alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin, and amylase and lipase. The central laboratory classified a finding as either abnormal or normal.
Time Frame: From Baseline until EOT (Week 24)
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Matching Placebo | Alitretinoin 30 mg
Number analyzed (Participants) | 9 | 24
Participants
  Triglycerides, BL normal, shift to abnormal | 0 | 2
  Triglycerides, BL abnormal, shift to abnormal | 0 | 0
  Total cholesterol BL normal, shift to abnormal | 1 | 1
  Total cholesterol BL abnormal, shift to abnormal | 0 | 1
  HDL cholesterol BL normal, shift to abnormal | 0 | 1
  HDL cholesterol BL abnormal, shift to abnormal | 0 | 0
  LDL cholesterol BL normal, shift to abnormal | 0 | 0
  LDL cholesterol BL abnormal, shift to abnormal | 0 | 1
  LDL/HDL ratio BL normal, shift to abnormal | 0 | 0
  LDL/HDL ratio BL abnormal, shift to abnormal | 0 | 0
  ALT BL normal, shift to abnormal | 0 | 0
  ALT BL abnormal, shift to abnormal | 0 | 0
  AST BL normal, shift to abnormal | 0 | 0
  AST BL abnormal, shift to abnormal | 0 | 0
  Bilirubin BL normal, shift to abnormal | 0 | 0
  Bilirubin BL abnormal, shift to abnormal | 0 | 0
  Amylase BL normal, shift to abnormal | 0 | 0
  Amylase BL abnormal, shift to abnormal | 0 | 0
  Lipase BL normal, shift to abnormal | 0 | 0
  Lipase BL abnormal, shift to abnormal | 0 | 0

14. Secondary Outcome: Mean Center for Epidemiological Studies Depression Scale (CES-D) Scores at Screening; Baseline; Weeks 4, 8, 12, 16, and 20; EOT (Week 24); and Safety Follow-up (Week 29)
Description: The CES-D scale is a short, self-report scale designed to measure depressive symptomatology in the general population. The CES-D consists of 20 questions. Participants were instructed to circle the number for each statement that best described how often they felt or behaved a particular way during the past week. The score was the sum of the weights of the 20 items. Responses range from 0 to 3 for each item (0=rarely or none of the time, 1=some or little of the time, 2=moderately or much of the time, 3=most or almost all the time). The CES-D score ranges from 0 to 60, with higher scores indicating greater depression. Participants with a CES-D score of 20 or higher were re-evaluated within 2 weeks. If a CES-D score of 20 or higher was confirmed on the second occasion, and if the score represents an increase over Baseline of 4 points or more, study treatment was interrupted and the participants were referred for psychiatric evaluation.
Time Frame: Screening; Baseline; Weeks 4, 8, 12, 16, and 20; EOT (Week 24); and safety follow-up (Week 29)
Population: Safety Population. Only participants available at the specified time points were analyzed (n=X, X).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Matching Placebo | Alitretinoin 30 mg
Number analyzed (Participants) | 9 | 24
Scores on a scale
  Screening, n=9, 23 | 7.2 (6.6) | 5.7 (4.7)
  Baseline, n=9, 24 | 7.0 (5.9) | 4.5 (5.9)
  Week 4, n=9, 20 | 5.0 (4.7) | 2.9 (3.5)
  Week 8, n=7, 20 | 2.7 (2.8) | 3.8 (6.7)
  Week 12, n=7, 17 | 4.0 (5.7) | 4.2 (6.6)
  Week 16, n=6, 16 | 3.8 (4.8) | 2.9 (5.5)
  Week 20, n=6, 14 | 4.0 (3.6) | 3.6 (5.2)
  End of Treatment, n=8, 20 | 7.4 (9.0) | 3.0 (5.4)
  Safety follow up, n=9, 22 | 4.4 (3.9) | 4.6 (6.7)

15. Secondary Outcome: Absolute Change From Baseline (BL) in CES-D Scores at Weeks 4, 8, 12, 16, and 20; EOT (Week 24); and Safety Follow-up (Week 29)
Description: The CES-D scale is a short, self-report scale designed to measure depressive symptomatology in the general population. The CES-D consists of 20 questions. Participants were instructed to circle the number for each statement that best described how often they felt or behaved a particular way during the past week. The score was the sum of the weights of the 20 items. Responses range from 0 to 3 for each item (0=rarely or none of the time, 1=some or little of the time, 2=moderately or much of the time, 3=most or almost all the time). The CES-D score ranges from 0 to 60, with higher scores indicating greater depression. Participants with a CES-D score of >=20 were re-evaluated within 2 weeks. If a CES-D score of >=20 was confirmed on the second occasion, and if the score represents an increase over BL of 4 points or more, study treatment was interrupted and the participants were referred for psychiatric evaluation. Change from BL is defined as the post-BL value minus the BL value.
Time Frame: Baseline; Weeks 4, 8, 12, 16, and 20; EOT (Week 24); and safety follow-up (Week 29)
Population: Safety Population. Only participants available at the specified time points were analyzed (n=X, X).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Matching Placebo | Alitretinoin 30 mg
Number analyzed (Participants) | 9 | 24
Scores on a scale
  Week 4, n=9, 20 | -2.0 (2.5) | -0.3 (2.4)
  Week 8, n=7, 20 | -2.3 (2.4) | 0.7 (7.5)
  Week 12, n=7, 17 | -1.0 (2.3) | 0.6 (5.4)
  Week 16, n=6, 16 | -2.0 (2.1) | -0.8 (4.7)
  Week 20, n=6, 14 | -1.8 (3.6) | 0.3 (4.7)
  End of Treatment, n=8, 20 | -0.5 (6.6) | -0.6 (4.7)
  Safety follow-up, n=9, 22 | -2.6 (3.9) | 0.1 (3.4)

16. Secondary Outcome: Mean Columbia Suicide Severity Rating Scale (CSSRS) Scores at Screening; Baseline; Weeks 4, 8, 12, 16, and 20; EOT (Week 24); and Safety Follow-up (Week 29)
Description: The assessment of suicidality was conducted using the CSSRS, a brief questionnaire designed to assess severity and change in suicidality using a semi-structured interview to probe participant responses. The suicidal ideation intensity total score was the sum of suicidal ideation severity rating scores for frequency, duration, controllability, deterrents, and reasons for ideation. For each item, each participant got an intensity score from 0(none) to 5(worst). Therefore, the suicidal ideation intensity total score range from 0 to 25, with a score of 0 given for no suicidal ideation. CSSRS scores were reported at Screening; Baseline; Week 4, 8, 12, 16, 20; EOT (Week 24);and safety follow-up (Week 29).
Time Frame: Screening; Baseline; Weeks 4, 8, 12, 16, and 20; EOT (Week 24), and safety follow-up (Week 29)
Population: Safety Population. Only participants available at the specified time points were analyzed (n=X, X).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Matching Placebo | Alitretinoin 30 mg
Number analyzed (Participants) | 9 | 24
Scores on a scale
  Screening, n=3, 10 | 0.0 (0.0) | 0.0 (0.0)
  Baseline, n=3, 10 | 0.0 (0.0) | 0.0 (0.0)
  Week 4, n=3, 09 | 0.0 (0.0) | 0.0 (0.0)
  Week 8, n=3, 09 | 0.0 (0.0) | 0.0 (0.0)
  Week 12, n=3, 07 | 0.0 (0.0) | 0.0 (0.0)
  Week 16, n=2, 07 | 0.0 (0.0) | 0.0 (0.0)
  Week 20, n=2, 6 | 0.0 (0.0) | 0.0 (0.0)
  End of Treatment, n=2, 7 | 0.0 (0.0) | 0.0 (0.0)
  Safety follow up, n=3, 9 | 0.0 (0.0) | 0.0 (0.0)

17. Secondary Outcome: Absolute Change From Baseline in the CSSRS Score at Weeks 4, 8, 12, 16, and 20; EOT (Week 24); and Safety Follow-up (Week 29)
Description: The assessment of suicidality was conducted using the CSSRS, a brief questionnaire designed to assess severity and change in suicidality using a semi-structured interview to probe participant responses. The suicidal ideation intensity total score was the sum of suicidal ideation severity rating scores for frequency, duration, controllability, deterrents, and reasons for ideation. For each item, each participant got an intensity score from 0(none) to 5(worst). Therefore, the suicidal ideation intensity total score range from 0 to 25, with a score of 0 given for no suicidal ideation. CSSRS scores were reported at Baseline; Week 4, 8, 12, 16, 20; EOT (Week 24); and safety follow-up (Week 29). Change from Baseline is defined as the value at the post-Baseline visit minus the Baseline value.
Time Frame: Baseline; Weeks 4, 8, 12, 16, and 20; EOT (Week 24); and safety follow-up (Week 29)
Population: Safety Population. Only participants available at the specified time points were analyzed (n=X, X).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Matching Placebo | Alitretinoin 30 mg
Number analyzed (Participants) | 9 | 24
Scores on a scale
  Week 4, n=3, 9 | 0.0 (0.0) | 0.0 (0.0)
  Week 8, n=3, 9 | 0.0 (0.0) | 0.0 (0.0)
  Week 12, n=3, 7 | 0.0 (0.0) | 0.0 (0.0)
  Week 16, n=2, 7 | 0.0 (0.0) | 0.0 (0.0)
  Week 20, n=2, 6 | 0.0 (0.0) | 0.0 (0.0)
  End of Treatment, n=2, 7 | 0.0 (0.0) | 0.0 (0.0)
  Safety follow-up, n=3, 9 | 0.0 (0.0) | 0.0 (0.0)

18. Secondary Outcome: Mean Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Screening, Baseline, and EOT (Week 24)
Description: SBP and DBP were assessed at Screening, Baseline, and EOT.
Time Frame: Screening, Baseline, and EOT (Week 24)
Population: Safety Population. Only participants available at the specified time points were analyzed (n=X, X).
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Matching Placebo | Alitretinoin 30 mg
Number analyzed (Participants) | 9 | 24
Millimeters of mercury (mmHg)
  SBP, Screening, n=9, 23 | 130.8 (13.7) | 131.3 (16.3)
  SBP, Baseline, n=9, 24 | 122.8 (14.0) | 126.3 (16.1)
  SBP, EOT, n=8, 20 | 122.4 (13.7) | 128.7 (21.4)
  DBP, Screening, n=9, 23 | 78.0 (10.7) | 79.7 (9.6)
  DBP, Baseline, n=9, 24 | 77.4 (12.2) | 79.1 (7.5)
  DBP, EOT, n=8, 20 | 76.0 (12.2) | 75.4 (10.5)

19. Secondary Outcome: Mean Heart Rate (HR) at Baseline, Screening, and EOT (Week 24)
Description: HR is defined as the rate at which the heart beats.
Time Frame: Screening, Baseline, and EOT (Week 24)
Population: Safety Population. Only participants available at the specified time points were analyzed (n=X, X).
Measure: Mean (Standard Deviation); unit: Beats per minute (bpm)
Arm/Group | Matching Placebo | Alitretinoin 30 mg
Number analyzed (Participants) | 9 | 24
Beats per minute (bpm)
  Screening, n=9, 23 | 68.3 (6.0) | 74.0 (7.3)
  Baseline, n=9, 24 | 72.3 (6.2) | 75.2 (8.8)
  EOT, n=8, 20 | 70.1 (6.6) | 74.7 (7.8)

20. Secondary Outcome: Mean Body Weight at Screening, Baseline ,and EOT (Week 24)
Description: Body weight was measured at Screening, Baseline, and EOT.
Time Frame: Screening, Baseline, and EOT (Week 24)
Population: Safety Population. Only participants available at the specified time points were analyzed (n=X, X).
Measure: Mean (Standard Deviation); unit: Kilograms (kg)
Arm/Group | Matching Placebo | Alitretinoin 30 mg
Number analyzed (Participants) | 9 | 24
Kilograms (kg)
  Screening, n=9, 24 | 89.3 (15.5) | 72.8 (12.6)
  Baseline, n=8, 24 | 89.6 (16.6) | 72.9 (12.9)
  EOT, n=8, 19 | 88.9 (16.5) | 73.8 (13.4)

21. Secondary Outcome: Change From Baseline in SBP and DBP at EOT (Week 24)
Description: Change from Baseline is defined as the value at EOT minus the Baseline value.
Time Frame: Baseline and EOT (Week 24)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Matching Placebo | Alitretinoin 30 mg
Number analyzed (Participants) | 8 | 20
mmHg
  SBP | 0.5 (12.5) | 0.7 (19.1)
  DBP | -0.5 (9.8) | -4.2 (9.8)

22. Secondary Outcome: Change From Baseline in Heart Rate at EOT (Week 24)
Description: HR is defined as the rate at which the heart beats. Change from Baseline is defined as the value at EOT minus the Baseline value.
Time Frame: Baseline and EOT (Week 24)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Matching Placebo | Alitretinoin 30 mg
Number analyzed (Participants) | 8 | 20
bpm | -3.1 (10.4) | -0.2 (10.2)

23. Secondary Outcome: Change From Baseline in Weight at EOT (Week 24)
Description: Change from Baseline is defined as the value at EOT minus the value at Baseline.
Time Frame: Baseline and EOT (Week 24)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Matching Placebo | Alitretinoin 30 mg
Number analyzed (Participants) | 7 | 19
kg | -0.8 (3.2) | -0.5 (1.4)

24. Secondary Outcome: Number of Participants With Normal/Abnormal Physical Status at Baseline With a Worst Post-Baseline Finding of Normal/Abnormal
Description: A physical examination for each participant was performed at Baseline and at EOT (Week 24). The primary investigator classified physical status as either normal or abnormal.
Time Frame: Baseline and EOT (Week 24)
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Matching Placebo | Alitretinoin 30 mg
Number analyzed (Participants) | 9 | 24
Participants
  Baseline normal, worst post-Baseline normal | 6 | 18
  Baseline normal, worst post-Baseline abnormal | 1 | 0
  Baseline abnormal, worst post-Baseline normal | 1 | 1
  Baseline abnormal, worst post-Baseline abnormal | 0 | 0

25. Secondary Outcome: Number of Participants With a Negative Serum Pregnancy Test at Screening; Baseline; Weeks 4, 8, 12, 16, and 20; EOT (Week 24); and Safety Follow-up (Week 29)
Description: Serum pregnancy tests were performed at each visit for females of childbearing potential.
Time Frame: Screening; Baseline; Weeks 4, 8, 12, 16, and 20; EOT (Week 24); safety follow-up (Week 29)
Population: Safety population. Only female participants were analysed for serum pregnancy test.
Measure: Number; unit: Participants
Arm/Group | Matching Placebo | Alitretinoin 30 mg
Number analyzed (Participants) | 5 | 14
Participants
  Screening | 4 | 7
  Baseline | 4 | 7
  Week 4 | 4 | 4
  Week 8 | 3 | 4
  Week 12 | 3 | 3
  Week 16 | 3 | 2
  Week 20 | 2 | 2
  EOT | 4 | 4
  Safety follow-up | 4 | 5

ADVERSE EVENTS:
Time Frame: AEs were recorded from date of randomization until the date of death from any cause, withdrawal from study or up to safety follow-up, whichever came first, assessed up to 29 weeks.
Description: SAEs and non-serious AEs were reported for members of the Safety Population, comprised of all randomized participants who received at least one dose of study medication.
Arm/Group | Matching Placebo | Alitretinoin 30 mg
Serious Adverse Events (participants affected / at risk) | 0/9 | 1/24
Other Adverse Events (participants affected / at risk) | 8/9 | 16/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Matching Placebo (N=9) | Alitretinoin 30 mg (N=24)
Dizziness (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Matching Placebo (N=9) | Alitretinoin 30 mg (N=24)
Nasopharyngitis (Infections and infestations) | 1 | 7
Bronchitis (Infections and infestations) | 1 | 1
Headache (Nervous system disorders) | 2 | 8
Cheilitis (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Blood triglycerides increased (Investigations) | 0 | 2
LDL/HDL ratio increased (Investigations) | 0 | 2
Low density lipoprotein increased (Investigations) | 0 | 2
Blood potassium increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 3
Gout (Metabolism and nutrition disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 2
Suicidal ideation (Psychiatric disorders) | 1 | 0
Granuloma annulare (Skin and subcutaneous tissue disorders) | 1 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hot flush (Vascular disorders) | 1 | 0
Discomfort (General disorders) | 1 | 0
Hepatic fibrosis (Hepatobiliary disorders) | 1 | 0
Allergy to arthropod bite (Immune system disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.